CLINICAL TRIAL: NCT00023205
Title: Literacy in Arthritis Management: A Randomized Controlled Clinical Trial of a Novel Education Intervention
Brief Title: Impact of Literacy Level on Patient Education and Health Among People With Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Matthew H. Liang, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: P60 AR47782 NIAMS-068; P60AR047782 (NIH)
Record Dates: First submitted 2001-08-29; First posted 2001-08-31 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Polyarthritis
Keywords: Arthritis; Health literacy; Patient education; Self-efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Individualized education (Experimental): Individualized education with materials written in plain language. Follow-up sessions/ phone contact as requested by the subject.
  Interventions: Behavioral: Interactive in-person arthritis education
- Standard care (Active Comparator): 1 session of education with provision of standard Arthritis Foundation materials.
  Interventions: Behavioral: 11th grade reading level arthritis materials

INTERVENTIONS:
Behavioral: 11th grade reading level arthritis materials
  Arms: Standard care
Behavioral: Interactive in-person arthritis education
  Arms: Individualized education

SUMMARY:
People with poor literacy may have worse health and less knowledge about how to manage their disease than patients at high reading levels. Patients with arthritis usually receive information on how to manage their disease that is written at an 11th grade reading level. The purpose of this study is to compare the health outcomes of patients with arthritis given either standard 11th grade level materials or interactive, in-person arthritis education along with materials written at a lower reading level.

DETAILED DESCRIPTION:
Patients with poor literacy report worse health and know less about managing their disease than patients with better literacy. This study will compare the disease outcomes of arthritis patients at three different reading levels who receive either standard arthritis materials written at an 11th grade reading level or an in-person, interactive, text-free session along with lower reading level materials. The study will determine the most effective methods of educating patients with poor literacy about their disease.

Patients with systemic inflammatory rheumatic conditions (rheumatoid arthritis, psoriatic arthritis, and seronegative polyarthritis) will be assessed and placed into one of three reading levels: 8th grade or lower; 9th to 11th grade; or 12th grade or higher. Patients from each reading level will be randomly assigned to one of two intervention groups. Group 1 will receive disease-specific material from the Arthritis Foundation written at an 11th grade reading level. Group 2 will receive plain language materials, an arthritis glossary, and a one-hour, in-person session with a study educator using interactive, text-free methods. The study educator will help the patient with reading-related problems either by study visit or by telephone for 6 months postsession.

All patients will receive a medication calendar. Patients will be followed for one year after the intervention and will be assessed for changes in health status, disease activity, communication with the physician, self-management of their arthritis, understanding of and adherence to prescribed treatment, and satisfaction with their intervention.

ELIGIBILITY:
Inclusion Criteria:

* Native English speaker
* Patient at the Rheumatology Clinic at Brigham and Women's Hospital, Boston, Massachusetts
* Diagnosis of rheumatoid arthritis, psoriatic arthritis, or seronegative polyarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2002-11; Primary Completion 2006-08 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | 6 months, 12 months
  self report of medication use on standard form
Self efficacy | 6 months and 12 months
  self report on self efficacy form
Satisfaction with medical care | 6 months and 12 months
  self report of satisfaction

SECONDARY OUTCOMES:
Heath Status | 6 months and 12 months
  Health Assessment questionaire
Mental Health | 6 months and 12 months
  SF-36 (5 items)
Understanding of medication | 6 months and 12 months
  open ended questionnaire of medication purpose
Perceived usefulness of materials | 6months and 12 months
  Interview
Appointment keeping | 6 and 12 months
  Clinical record

OTHER OUTCOMES:
Literacy-related problems encountered in management | 6 months and 12 months
  Interview

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Liang, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Weiss BD, Hart G, McGee DL, D'Estelle S. Health status of illiterate adults: relation between literacy and health status among persons with low literacy skills. J Am Board Fam Pract. 1992 May-Jun;5(3):257-64. PMID 1580173
- [Background] Kitsch I, A. Jungeblut, L. Jenkins, and A. Kolstad. Adult Literacy in America: A First Look at the Results of the National Adult Literacy Survey. Washington, DC: National Center for Education Statistics, US Department of Education; 1993.